CLINICAL TRIAL: NCT05487092
Title: Letrozole in Preventing Recurrence of Endometrioma Following Laparoscopic Ovarian Cystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Pamela Youde Nethersole Eastern Hospital (Other); The Queen Elizabeth Hospital (Other); Kwong Wah Hospital (Other); Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UW21-556
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Endometriotic Cyst of Ovary
Keywords: endometriotic cyst; recurrence; letrozole; combined oral contraceptive pills
MeSH Terms: conditions — Endometriosis; Recurrence | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Letrozole (Experimental): They will be given letrozole 2.5mg daily on top of combined oral contraceptive (COC) pills (Microgynon 30, which contains 30mcg ethinyloestradiol and 150 mcg levonorgestrel) orally for 6 months after laparoscopic ovarian cystectomy, followed by COC pills alone subsequently as routine
  Interventions: Drug: Letrozole
- Standard treatment (Placebo Comparator): They will be given placebo tablets (which will be identical to letrozole) on top of COC pills (Microgynon 30, which contains 30mcg ethinyloestradiol and 150 mcg levonorgestrel) orally for 6 months after laparoscopic ovarian cystectomy, followed by COC pills alone subsequently
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Letrozole — Letrozole 2.5mg daily for 6 months
  Arms: Letrozole
Other: Placebo — Placebo
  Arms: Standard treatment

SUMMARY:
Endometriosis is a chronic inflammatory disease that affects approximately 10-15% of women of reproductive age. Symptoms include dysmenorrhoea, chronic pelvic pain, dyspareunia and infertility. Removal of the endometriotic cyst (chocolate cyst) by surgery is a well-established treatment for symptomatic relief. However, recurrence of endometriotic cyst after surgical removal of the cyst is up to 30-50% after ovarian surgery. Oral contraceptive pills for 18-24 months after the surgery is widely used as a postoperative hormonal therapy because it has been shown to reduce the chance of recurrence of the endometriotic cyst, but recurrence is still high even after taking oral contraceptive pills.

Letrozole is an aromatase inhibitor. There are some preliminary reports that letrozole can cause shrinkage of endometriotic cysts and improve endometriosis-related pelvic pain by reducing oestrogen level, inflammation and stem cell recruitment that may be important in recurrence of endometriotic cyst. This is a randomized double-blinded placebo-controlled trial. The aim of this study is to assess whether taking letrozole in addition to oral contraceptive pills in the first 6 months after laparoscopic surgery (key-hole surgery) to remove the endometriotic cyst can reduce the risk of recurrence compared to oral contraceptive pills alone. The study also involves laboratory parts from a small portion of the endometriotic cyst specimens (removed during laparoscopy ovarian cystectomy) and endometrial biopsy (if the patient agrees) to assess the role of stem cells in the pathogenesis of endometriotic cysts.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years old
* Scheduled to have laparoscopic ovarian cystectomy
* Unilateral or bilateral endometrioma on pre-operative ultrasound and confirmed by histology

Exclusion Criteria:

* Use of long-acting hormonal therapy in the 3 months before inclusion in the study
* Histological report of laparoscopic ovarian cystectomy showed atypical endometrioma
* Complex surgery including resection of deep infiltrating disease, bowel resection or hysterectomy
* Incomplete excision of endometrioma/ incision or drainage rather than ovarian cystectomy
* Suspicion of malignancy
* Contraindications to combined oral contraceptive pills, including: uncontrolled hypertension (systolic > 160mmHg or diastolic > 100mmHg), diabetes with retinopathy/ nephropathy/ neuropathy, current or past history of venous thromboembolism, ischemic heart disease, history of cerebrovascular accident, migraine with aura, severe liver disease, oestrogen-sensitive cancers, undiagnosed abnormal uterine bleeding, smokers (> 15 cigarettes/day) aged 35 years or above, or having body mass index >=35 kg/m2
* Planning to get pregnant in the coming 1 year
* Refusal to join the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 194 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence of endometrioma | 12 months
  the presence of ovarian cysts with the typical sonographic criteria of endometriomas and a diameter of ≥30 mm after previous complete ovarian cystectomy, to be measured by a transvaginal or transrectal ultrasound transducer

SECONDARY OUTCOMES:
Endometriosis Health Profile Questionnaire (EHP-30) score | 6 months, 12 months, 24 months
  a validated disease-specific health related quality of life patient self-reported scale for endometriosis used to measure the effects that endometriosis can have on the women's lives and the effectiveness of medical and surgical therapies for endometriosis on their quality of life
Non-menstrual pelvic pain (chronic pelvic pain, deep dyspareunia) and dysmenorrhoea measured by a 10cm visual analogue pain scale (VAS) | 6 months, 12 months, 24 months
  0-100
Menstrual regularity | 6 months, 12 months, 24 months
  menstrual chart
Use of additional analgesics | 6 months, 12 months, 24 months
Side effects/ adverse events | 6 months, 12 months, 24 months
  Number of women with side effects/ adverse events
Need for further surgery for endometriosis | 6 months, 12 months, 24 months
  Number of women who required further surgery for endometriosis

CONTACTS AND LOCATIONS:
Locations (5):
- Hong Kong (5):
  - Queen Mary Hospital, Hong Kong
  - Kwong Wah Hospital, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No